CLINICAL TRIAL: NCT07408050
Title: A Study on the Reconstruction of Complex Ureteral Stenosis Utilizing Preputial Grafts.
Brief Title: An Investigation Into the Application of Preputial Grafts for the Reconstruction of Complex Ureteral Strictures
Acronym: PGU20240101
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ruibao chen (Other)
Responsible Party: Sponsor-Investigator, Ruibao chen, Principal Investigator, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TJ-IRB202505033; MR-42-25-056915 (Registry Identifier: China National Medical Research Registration and Filing Information System)
Record Dates: First submitted 2026-01-27; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Ureteral Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with complex ureteral stenosis undergoing PGU surgery (Experimental): After enrolling patients with complex ureteral stenosis, PGU surgery was performed, and postoperative follow-up was conducted to assess complications, renal hydronephrosis, and renal function recovery.
  Interventions: Procedure: Preputial graft ureteroplasty

INTERVENTIONS:
Procedure: Preputial graft ureteroplasty — Reconstruction of complex ureteral stenosis using preputial graft

SUMMARY:
Complex ureteral stricture refers to a ureteral lumen stenosis lesion that cannot be directly treated with the traditional end-to-end anastomosis. In recent years, its incidence has shown a gradual upward trend, and it has long been a major clinical challenge for urological surgeons. Because it is difficult to achieve tension-free anastomosis after direct resection of the strictured segment, which can easily lead to the failure of stricture repair surgery, simple ureteral stricture segment resection combined with end-to-end anastomosis is generally not recommended for the treatment of such diseases.

In general, clinicians need to select alternative materials for ureteral reconstruction, such as Boari flap, appendix, intestinal tract, and oral mucosa, to achieve the surgical effect of tension-free anastomosis. However, in some complex clinical cases, if Boari flap, appendix, intestinal tract or oral mucosa cannot be used for surgery, or if patients refuse to accept oral mucosa, intestinal mucosa and other tissues for ureteral repair, are there any other alternative schemes with high safety and minimal invasiveness available for ureteral reconstruction in clinical practice? Thus, it is of great clinical significance to develop safe, effective and innovative surgical techniques for ureteral reconstruction. Circumcision is a surgical procedure with a long history and wide application, and the prepuce removed during the operation is usually treated as medical waste. Our research team has previously performed a large number of surgeries using prepuce to repair the urethra. Clinical results have shown that free prepuce has the advantages of easy survival, convenient harvesting and minimal invasiveness, making it an ideal graft material for urinary tract repair and reconstruction.

At present, there have been case reports on ureteral reconstruction using prepuce abroad. Based on our team's previous research experience in the fields of urethral reconstruction and ureteral reconstruction, the investigators intend to carry out relevant research on ureteral reconstruction with free preputial grafts, aiming to obtain convincing clinical data and provide a more minimally invasive and safer new treatment option for the repair and reconstruction of complex ureteral strictures.

ELIGIBILITY:
Inclusion Criteria

* Male patients over 18 years of age.
* Preoperative assessment confirming complex ureteral strictures, characterized by ureteral luminal stenosis that cannot be addressed via conventional end-to-end anastomosis. Patients were deemed ineligible for existing surgical. interventions such as pyeloureteroplasty, ureteral end-to-end anastomosis, and ureteroneocystostomy.
* Ability to undergo minimally invasive laparoscopic surgery for ureteral stricture repair.
* Presence of redundant prepuce or availability of an inner preputial flap for graft harvesting.
* Capacity for independent decision-making and willingness to voluntarily sign the informed consent form for study participation.

Exclusion Criteria

* Presence of surgical contraindications.
* History of abdominal radiotherapy.
* Ureteral strictures resulting from malignant tumors.
* An Eastern Cooperative Oncology Group (ECOG) performance status score greater than 2.
* Poor compliance or other exclusion criteria as determined by the investigators.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-02-05 (Estimated); Primary Completion 2031-01-01 (Estimated); Study Completion 2032-01-01 (Estimated)

PRIMARY OUTCOMES:
Ureteral patency | From surgery to 6 months after surgery
  The alteration in eGFR, denoted as ΔeGFR, was employed to evaluate changes in renal function. The calculation for ΔeGFR is as follows: ΔeGFR = (postoperative eGFR - preoperative eGFR) / preoperative eGFR. Renal ultrasound, computed tomography (CT), and magnetic resonance urography (MRU) are utilized to measure the anteroposterior diameter (APD) and indirectly assess ureteral patency.

IPD SHARING:
Plan to Share IPD: Yes
International Committee of Medical Journal Editors
Supporting Information: Study Protocol, SAP, CSR
Time Frame: From 20260206 to 20310101
Access Criteria: ICMJE will be able to access the IPD and supporting information. They will be able to access Study Protocol,Statistical Analysis Plan, and Clinical Study Report.
URL: https://www.medicalresearch.org.cn/clinicalResearch/researchMain